CLINICAL TRIAL: NCT05295628
Title: A Prospective, Randomized, Multicenter Evaluation of the Safety and Effectiveness of the EMBLOK Embolic Protection System During Transcatheter Aortic Valve Replacement
Brief Title: Evaluation of Safety and Effectiveness of the EMBLOK EPS During TAVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emblok, Inc. (Industry)
Collaborators: Yale Cardiovascular Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLP 001-2021
Record Dates: First submitted 2022-02-21; First posted 2022-03-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 532 subjects undergoing TAVR at up to 30 investigational sites in the United States.
  Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects (up to 60 subjects total), who will not be randomized but will receive the EMBLOK EPS during TAVR.
  In the randomized cohort, up to 422 subjects meeting eligibility criteria will be randomized 1:1 (stratified by operative risk and study site) to one of two treatment arms:
  1. Intervention - EMBLOK EPS during TAVR
  2. Control - SENTINEL CPS during TAVR
  In addition, a nested registry will enroll up to 50 subjects who meet clinical eligibility criteria and are anatomically suitable for the EMBLOK EPS, but whose anatomy precludes the use of the SENTINEL CPS.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blind study. The following individuals will be blinded to the subject's treatment allocation:
  * The subject and his or her family members
  * Site personnel administering neurological evaluations
  * Pathology Core Laboratory personnel performing debris analyses
  Un-blinding will occur only after the database has been locked for the analysis of the primary endpoint or to protect subject rights, welfare, or well-being at the request of the DMC. A site investigator may also reveal treatment allocation to an individual subject if deemed necessary due to complication or injury.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EMBLOK™ Embolic Protection System (Experimental): Device Description:
  The EMBLOK™ Embolic Protection System ("EMBLOK EPS") is a sterile, single use system designed to capture and remove debris (e.g., thrombus, calcium, atheroma) dislodged during transcatheter aortic valve replacement (TAVR) procedures. The device is currently for investigational use only.
  When Device Will Be Used:
  Roll-in: Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects, who will not be randomized but will receive the EMBLOK EPS during TAVR.
  Randomized: Up to 422 subjects meeting eligibility criteria will be randomized 1:1. The experimental "intervention" arm is utilizing EMBLOK EPS during TAVR (up to 211 subjects).
  Nested registry: Up to 50 subjects who meet clinical eligibility criteria and are anatomically suitable for the EMBLOK EPS, but whose anatomy precludes the use of the SENTINEL CPS.
  Interventions: Device: EMBLOK™ Embolic Protection System ("EMBLOK EPS")
- SENTINEL™ Cerebral Protection System (Active Comparator): Device Description:
  The control comparator is the commercially-available SENTINEL™ Cerebral Protection System ("SENTINEL CPS") (Boston Scientific Corp., Marlborough, MA, US), a dual-filter protection device designed to capture and remove debris dislodged during TAVR procedures.
  The SENTINEL CPS is indicated for use as an embolic protection device to capture and remove thrombus/debris while performing TAVR procedures. The diameters of the arteries at the site of filter placement should be between 9.0 mm - 15.0 mm for the brachiocephalic and 6.5 mm - 10.0 mm in the left common carotid.
  When Device Will Be Used:
  In the randomized cohort, up to 422 subjects meeting eligibility criteria will be randomized 1:1 (stratified by operative risk and study site). The active comparator "control" arm is utilizing SENTINEL CPS during TAVR (up to 211 subjects).
  Interventions: Device: SENTINEL™ Cerebral Protection System

INTERVENTIONS:
Device: EMBLOK™ Embolic Protection System ("EMBLOK EPS") — The EMBLOK EPS is intended to capture and remove thrombus/debris while performing transcatheter aortic valve replacement procedures.
  Arms: EMBLOK™ Embolic Protection System
Device: SENTINEL™ Cerebral Protection System — The SENTINEL CPS is intended to capture and remove thrombus/debris while performing transcatheter aortic valve replacement procedures.
  Arms: SENTINEL™ Cerebral Protection System

SUMMARY:
The objective of the study is to evaluate the safety, effectiveness, and performance of the EMBLOK EPS during TAVR by randomized comparison with a commercially available embolic protection device. The targeted study population consists of patients meeting FDA-approved indications for TAVR with commercially available transcatheter heart valve systems.

This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 532 subjects undergoing TAVR at up to 30 investigational sites in the United States. All subjects will undergo clinical follow-up (including detailed neurological assessments) in-hospital and at 30 days.

DETAILED DESCRIPTION:
Embolic stroke remains a major complication for TAVR, resulting in a two-fold increase in 1-year mortality. Embolic protection devices have been developed to filter embolic debris during the procedure, potentially reducing the occurrence of neurologic events associated with TAVR. The EMBLOK EPS may improve on currently available devices by capturing and retrieving debris directed toward all 3 cerebral vessels in the aortic arch as well as the descending aorta.

The objective of the study is to evaluate the safety, effectiveness, and performance of the EMBLOK EPS during TAVR by randomized comparison with a commercially available embolic protection device. With this comparator device, the left subclavian artery and descending aorta are not protected.

The targeted study population consists of patients meeting FDA-approved indications for TAVR with commercially available transcatheter heart valve systems.

This prospective, multicenter, single-blind, randomized controlled trial will enroll up to a total of 532 subjects undergoing TAVR at up to 30 investigational sites in the United States.

Prior to enrollment of the first randomized subject at each site, each site will enroll 2 Roll-In subjects (up to 60 subjects total), who will not be randomized but will receive the EMBLOK EPS during TAVR.

In the randomized cohort, up to 422 subjects meeting eligibility criteria will be randomized 1:1 (stratified by operative risk and study site) to one of two treatment arms:

1. Intervention - EMBLOK EPS during TAVR
2. Control - SENTINEL CPS during TAVR

In addition, a nested registry will enroll up to 50 subjects who meet clinical eligibility criteria and are anatomically suitable for the EMBLOK EPS, but whose anatomy precludes the use of the SENTINEL CPS.

All subjects will undergo clinical follow-up (including detailed neurological assessments) in-hospital and at 30 days.

ELIGIBILITY:
Clinical Eligibility Criteria:

Clinical Inclusion Criteria:

Subjects must meet ALL the following criteria to be eligible for participation in the study:

1. Subject is between 18 and 90 years of age.
2. Subject meets FDA approved indications for TAVR procedure on a native aortic valve using an iliofemoral approach with a commercially approved transcatheter heart valve.
3. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 48 hours prior to the index study procedure.
4. Subject agrees to comply with all protocol-specified procedures and assessments.
5. Subject or subject's legal representative signs an IRB approved informed consent form prior to study participation.

Clinical Exclusion Criteria:

Subjects will be excluded if ANY of the following criteria apply:

1. Subjects with a previously implanted aortic or mitral valve bioprosthesis
2. Subjects with hepatic failure (Child-Pugh class C).
3. Subjects with hypercoagulable states that cannot be corrected by additional periprocedural heparin.
4. Subjects who have a planned treatment with any other investigational device or procedure during the study period.
5. Subjects planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVR procedure or within 10 days prior to the TAVR procedure. NOTE: Diagnostic cardiac catheterization is permitted within 10 days prior to the TAVR procedure.
6. Subject has experienced an acute myocardial infarction (World Health Organization [WHO] criteria) within 30 days of the planned index procedure.
7. Subject requires an urgent or emergent TAVR procedure.
8. Subjects with renal failure (estimated Glomerular Filtration Rate [eGFR] < 30 mL/min by the Modification of Diet in Renal Disease [MDRD] formula).
9. Subject has documented history of stroke or transient ischemic attack within prior 6 months, or any prior stroke with a permanent major disability or deficit.
10. Subject has an ejection fraction of 30% or less.
11. Subject has a sensitivity to contrast media that cannot be adequately pre-treated.
12. Subject has known allergy or hypersensitivity to any embolic protection device materials (e.g., nickel-titanium) or allergy to intravascular contrast agents that cannot be pre-medicated
13. Subject has active endocarditis or an ongoing systemic infection defined as fever with temperature > 38°C and/ or white blood cell > 15,000 IU.
14. Subjects undergoing therapeutic thrombolysis.
15. Subject has history of bleeding diathesis or a coagulopathy or contraindications to anticoagulation and antiplatelet therapy.
16. Subject is known or suspected to be pregnant, or is lactating.
17. Subject is currently participating in another drug or device clinical study, or has other medical illnesses that may cause the subject to be non-compliant with the protocol or confound the data interpretation.

Anatomic Eligibility Criteria:

General Anatomic Exclusion Criteria:

Subjects meeting any of the following criteria will not be eligible for participation in the study:

1. Non-iliofemoral approach for is required for the TAVR system (e.g., trans-axillary, trans-subclavian, trans-brachiocephalic, trans-carotid, trans-apical or trans-aortic access for TAVR is required).
2. Subject peripheral anatomy is not compatible with contralateral iliofemoral access with an 11 French catheter (e.g., due to excessive tortuosity, stenosis, ectasia, dissection, or aneurysm).
3. Ascending aorta length (from the site of filter placement to the aortic root) less than 7.5 cm.
4. Diameter of the aorta at the intended site of Emblok filter deployment proximal to the brachiocephalic artery ostium is less than 25 mm or greater than 40 mm.
5. Subjects with severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery sheath vascular access.
6. Subjects in whom the aortic arch is heavily calcified, severely atheromatous, or severely tortuous.

Additional Anatomic Exclusion Criteria:

Subjects with any of the following criteria will be excluded from participation in the Randomized Cohort, but are eligible for participation in the Roll-In and Nested Registry cohorts (provided they meet all other eligibility criteria):

1. Diameters of the arteries at the site of filter placement are < 9 or > 15 mm for the brachiocephalic artery or < 6.5 or >10 mm in the left common carotid.
2. Brachiocephalic or carotid vessel with excessive tortuosity.
3. Compromised blood flow to the right upper extremity, or other conditions that would preclude 6 Fr radial or brachial vascular access (e.g., excessive tortuosity)
4. Arterial stenosis >70% in either the left common carotid artery or the brachiocephalic artery.
5. Brachiocephalic or left carotid artery reveals significant stenosis, ectasia, dissection, or aneurysm at the aortic ostium or within 3 cm of the aortic ostium.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite of all-cause mortality, all stroke (disabling or non-disabling) and transient ischemic attack (TIA), and Acute Kidney Injury Stage 2 or 3 (including renal replacement therapy), according to VARC-2 definitions | Evaluated at 30-day post-procedure (TAVR) follow-up visit
  The primary safety and efficacy endpoint is combined safety and efficacy at 30 days, defined as a composite of the following VARC-2 defined components:
  * All-cause mortality
  * All stroke (disabling or non-disabling) and transient ischemic attack (TIA)
  * Acute Kidney Injury Stage 2 or 3 (including renal replacement therapy)
Debris capture, defined as the average number of captured particles ≥150 µm in diameter, as assessed by independent histologic analysis | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  The co-primary filtration efficacy endpoint is debris capture, defined as the average number of captured particles ≥150 μm in diameter, as assessed by independent histologic analysis.

SECONDARY OUTCOMES:
Incidence of the composite of all-cause mortality, all stroke (disabling or non-disabling) and transient ischemic attack (TIA), and Acute Kidney Injury Stage 2 or 3 (including renal replacement therapy), according to VARC-2 definitions | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up until 7 days post procedure, which ever occurs first.
  Combined safety and efficacy is defined as a composite of the following VARC-2 defined components, evaluated post-procedure and in-hospital:
  * All-cause mortality
  * All stroke (disabling and non-disabling) and transient ischemic attack (TIA)
  * Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
Incidence of all-cause mortality (VARC-2 defined), subclassified as cardiovascular or non-cardiovascular mortality | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up until 7 days post procedure, which ever occurs first.
  Mortality (VARC-2 defined), evaluated in-hospital, defined as:
  • All-cause mortality
  * Cardiovascular mortality
  * Non-cardiovascular mortality
Incidence of stroke (sub-classified as ischemic, hemorrhagic, or undetermined, and as disabling or non-disabling) and TIA, according to VARC-2 and NeuroARC definitions | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Neurological Events (VARC-2 and NeuroARC defined)
  * Stroke (sub-classified as ischemic, hemorrhagic, or undetermined, and as disabling or non-disabling)
  * TIA
Incidence of acute kidney injury (AKIN classification), subclassified as stage 1, 2, or 3 | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Acute Kidney Injury (AKIN Classification)
  * AKI Stage 1
  * AKI Stage 2
  * AKI Stage 3
Incidence of life-threatening or disabling bleeding and major bleeding (VARC-2 defined) | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Bleeding Complications (VARC-2 defined)
  * Life-threatening or disabling bleeding
  * Major bleeding
Incidence of major vascular complications | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  Vascular Complications
  • Major vascular complications
Incidence of the composite of all stroke (disabling or non-disabling) and transient ischemic attack (TIA), and Acute Kidney Injury Stage 2 or 3 (including renal replacement therapy), and systemic embolization | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up until 7 days post procedure, which ever occurs first.
  Major adverse embolic events (MAEE)
  MAEE will be reported as a composite and components [evaluated post-procedure and in-hospital]:
  * All stroke (disabling and non-disabling) or TIA
  * Acute kidney injury (Stage 2 or 3, including RRT)
  * Systemic embolization
Prevalence of captured embolic debris, as assessed by an independent Pathology Core Laboratory | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Gross and histologic evaluation of captured embolic debris, including particle presence, will be assessed by an independent Pathology Core Laboratory.
Number of captured particles, as assessed by an independent Pathology Core Laboratory | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Gross and histologic evaluation of captured embolic debris, including particle count, will be assessed by an independent Pathology Core Laboratory.
Diameter of captured particles (in mm), as assessed by an independent Pathology Core Laboratory | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Gross and histologic evaluation of captured embolic debris, including particle size, will be assessed by an independent Pathology Core Laboratory.
Material composition of captured particles, as assessed by an independent Pathology Core Laboratory | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Gross and histologic evaluation of captured embolic debris, including particle composition, will be assessed by an independent Pathology Core Laboratory.
Neurocognitive Measures: NIHSS assessment | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  NIHSS worsening, defined as an increase of 2 or more points from baseline, assessed on the National Institutes of Health Stroke Scale (scores range from 0 to 42; higher scores mean worse outcome).
Neurocognitive Measures: MoCA assessment | Evaluated immediately after the intervention/procedure, up until discharge from hospital or up to 7 days post-procedure, and at the 30 day follow-up visit.
  MoCA worsening, defined as a decrease of 2 or more points from baseline, assessed on the Montreal Cognitive Assessment (scores range from 0 to 30; higher scores mean better outcomes).
Rate of successful device delivery to the site of filter placement and successful deployment of the device | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Secondary Performance Endpoint:
  • Successful device deployment, defined as ability to successfully deliver the device to the site of filter placement and successfully deploy the device.
Rate of successful device positioning followed by maintenance of positioning for the duration of the TAVR procedure, as assessed by an independent Angiographic Core Laboratory | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Secondary Performance Endpoint:
  • Successful device positioning, defined as ability to position the device and to maintain the device in place for the duration of the TAVR procedure (as assessed by an independent Angiographic Core Laboratory)
Rate of successful retrieval of the intact device | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Secondary Performance Endpoint:
  • Successful device retrieval, defined as ability to retrieve the device intact
Rate of successful deployment, positioning, and retrieval of the device | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Secondary Performance Endpoint:
  • Device success, defined as successful deployment, positioning and retrieval
Rate of successful deployment, positioning, and retrieval of the device without embolic protection device-related serious adverse events | Evaluated at the time of the TAVR procedure (during the intervention/procedure)
  Secondary Performance Endpoint:
  • Procedure success, defined as device success in the absence of in-hospital embolic protection device-related serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hemal Gada, MD, Principal Investigator — Heart and Vascular Institute, UPMC Pinnacle
Locations (23):
- United States (23):
  - Dignity Health Chandler Regional Medical Center, Chandler, Arizona
  - St Joseph's Providence, Orange, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Ascension Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - University of Washington School of Medicine Barnes Jewish Hospital, St Louis, Missouri
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Scott and White The Heart Hospital Plano- Baylor Institute of Research, Plano, Texas
  - Methodist Hospital, San Antonio, Texas
  - Sentra Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No